CLINICAL TRIAL: NCT01045265
Title: Study to Determine the Concentrations of Raltegravir in Semen, the Seminal to Plasma Ratio of Raltegravir and the Variability in Seminal to Plasma Ratios Over the Raltegravir Dosing Period.
Brief Title: Concentrations of Raltegravir in the Semen of HIV-Infected Men
Status: Completed | Type: Observational
Sponsor: Canadian Immunodeficiency Research Collaborative (Other)
Responsible Party: Sponsor
Other Study IDs: MISP35369
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Results first posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Raltegravir treated men: Single group study of seminal plasma pharmacokinetics of raltegravir in men receiving chronic raltegravir therapy
  Interventions: Other: Seminal plasma pharmacokinetics

INTERVENTIONS:
Other: Seminal plasma pharmacokinetics — Measure semen sample concentrations, obtain semen to plasma ratios across the dosing interval, the area under the concentration time curve of raltegravir in semen, the variability in penetration of raltegravir into the seminal compartment over the dosing period.

SUMMARY:
The objective of this study is to determine if concentrations of raltegravir in semen exceed the 50% and 95% inhibitory concentrations of HIV during the dose interval.

The secondary objective is to determine the extend of raltegravir penetration into semen by obtaining semen to plasma ratios across the dosing interval, to determine the area under the concentration time curve of raltegravir in semen, and to determine the variability in the penetration of raltegravir into the seminal compartment over the dosing period.

DETAILED DESCRIPTION:
The patient population will consist of 12 male HIV-positive patients who have been receiving stable antiretroviral therapy that includes raltegravir for a minimum of three months. Patients will be enrolled from one clinic in downtown Toronto and a hospital affiliated HIV specialty clinic in Ottawa, Ontario. Eligible patients will have evidence of full virologic suppression (HIV viral load < 50 copies/mL) at least one month prior to enrollment in the study. No changes will be made to the patients antiretroviral therapy during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected male
* 18 years old or older
* on raltegravir twice daily as part of their antiretroviral regimen for at least 3 months prior to screening
* viral load < 50 copies/mL at least one month prior to enrolling
* able to read, understand and sign a written informed consent prior to initiation of the study
* medically stable at the time of the study, with no evidence of acute illness

Exclusion Criteria:

* having difficulty adhering to current antiretroviral therapy
* patient is expected to have difficulties adhering with study protocol
* patients with malignancy, or acute renal or liver disease
* patient with active AIDS-defining illness
* patient with any medical, psychiatric or other circumstance that may impede the provision of informed consent
* patient with any of the following abnormalities at the time of screening:
* hemoglobin < 85 g/L
* absolute neutrophil count < 1000 cells/uL
* platelet count < 50,000 cells/ microleter (uL)
* aspartate aminotransferase (AST), alanine transaminase (ALT) or total bilirubin > 3 times the upper limit of normal
* serum creatinine > 1.5 times upper limit of normal
* patient receiving concomitant therapy with rifampin or St. John's wort

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 12 HIV-positive males
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2009-12; Primary Completion 2011-09 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mona Loutfy, MD, MPH, Principal Investigator — Maple Leaf Medical Research; Tony Antoniou, Principal Investigator — Unity Health Toronto
Locations (2):
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Canadian Immunodeficiency Research Collaborative, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Men on Raltegravir: HIV-infected men on chronic therapy with raltegravir 400 mg per day as part of antiretroviral therapy regimen.
Period: Overall Study
Arm/Group | Men on Raltegravir
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The median age and baseline CD4+ T-cell count of the study participants were 48 years (IQR 42-53) and 450 cells/mm3 (IQR 289-585).
Groups:
- Men on Raltegravir: Measuring semen samples: Measure semen sample concentrations, obtain semen to plasma ratios across the dosing interval, the area under the concentration time curve of raltegravir in semen, the variability in penetration of raltegravir into the seminal compartment over the dosing period.
Arm/Group | Men on Raltegravir
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [42 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Region of Enrollment [Number; unit: participants]
  Canada | 16
CD4 Count [Median (Inter-Quartile Range); unit: cells/mm^3] | 450 [289 to 585]

OUTCOME MEASURES:

1. Primary Outcome: Seminal Concentrations of Raltegravir.
Description: Determine if concentrations of raltegravir in semen exceed the 50% and 95% inhibitory concentrations of HIV during the dosing interval.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: mg/l
Groups:
- 16 Male HIV-positive Patients: Measuring semen samples: Measure semen sample concentrations, obtain semen to plasma ratios across the dosing interval, the area under the concentration time curve of raltegravir in semen, the variability in penetration of raltegravir into the seminal compartment over the dosing period.
Arm/Group | 16 Male HIV-positive Patients
Number analyzed (Participants) | 16
mg/l
  C-min | 0.18 [0.13 to 0.24]
  C-max | 1.91 [1.46 to 4.33]

2. Secondary Outcome: Semen to Plasma Raltegravir Concentrations
Description: Determine the extent of raltegravir penetration into semen by obtaining semen to plasma ratios across the dosing interval.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | 16 Male HIV-positive Patients
Number analyzed (Participants) | 16
ratio | 3.25 [1.46 to 5.37]

3. Secondary Outcome: Seminal Distribution of Raltegravir
Description: Determine the area under the concentration time curve of raltegravir in semen.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: h mg/l
Arm/Group | 16 Male HIV-positive Patients
Number analyzed (Participants) | 16
h mg/l | 6.83 [5.24 to 13.47]

4. Secondary Outcome: Semen to Plasma Distribution of Raltegravir
Description: Determine the variability in the penetration of raltegravir into the seminal compartment over the raltegravir dosing period.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | 16 Male HIV-positive Patients
Number analyzed (Participants) | 16
ratio | 2.26 [1.05 to 4.45]

ADVERSE EVENTS:
Time Frame: collected over 1.5 years
Groups:
- Men on Raltegravir: HIV-infected men receiving chronic therapy with raltegravir 400 mg per day as part of antiretroviral regimen.
Arm/Group | Men on Raltegravir
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days